CLINICAL TRIAL: NCT04629456
Title: Neuromuscular Electric Stimulation and Exercises Effect on Functional Exercise Performance and Quality of Life in Cases of Liver Cirrhosis
Brief Title: Physical Therapy for Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manal k. youssef, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T. REC/012/002609
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: liver cirrhosis; exercises; neuromuscular electric stimulation; exercise capacity; quality of life
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Liver Cirrhosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): A total of eight electrodes were placed on the quadriceps femoris muscles (four on each leg): two on the vastus medialis, one on the rectus femoris muscle, and one on the vastus lateralis muscle. The stimulation protocol of the NMES consisted of a symmetrical biphasic square pulse at 75 Hz, a duty cycle of 6 seconds (sec.) on and 29 sec. off, a pulse time of 410 sec. during a session lasting 20 min. The intensity was increased to maximum individual toleration. The muscle contractions were visible and palpable.
  Interventions: Other: neuromuscular electric stimulation
- Group 2 (Experimental): The chair-seated exercises were used in the early stages of the program because the participants were frail adults. Repetitions of toe raises, heel raises, knee lifts, knee extensions, and others were performed while seated on a chair. Hip flexions, lateral leg raises, and repetitions of other exercises were performed standing upright behind the chair and holding the back of the chair for stability. To strengthen lower extremities, a fixed weight was placed on the ankle while participants performed strengthening exercises. Weights of 0.50, 0.75, 1.00, and 1.50 kg were used in accordance with each participant's strength level as the resistance progressively increased. The exercises performed using these ankle weights included seated knee flexion and extension and standing knee flexion and extensions. Exercises using a resistance band: Resistance bands were used to strengthen lower body. Lower body exercises included leg extension and hip flexion(24).
  Interventions: Other: Exercises

INTERVENTIONS:
Other: neuromuscular electric stimulation — A total of eight electrodes were placed on the quadriceps femoris muscles (four on each leg): two on the vastus medialis, one on the rectus femoris muscle, and one on the vastus lateralis muscle. The stimulation protocol of the NMES consisted of a symmetrical biphasic square pulse at 75 Hz, a duty cycle of 6 seconds (sec.) on and 29 sec. off, a pulse time of 410 sec. during a session lasting 20 min. The intensity was increased to maximum individual toleration. The muscle contractions were visible and palpable.
  Arms: group 1
Other: Exercises — The chair-seated exercises were used in the early stages of the program because the participants were frail adults. Repetitions of toe raises, heel raises, knee lifts, knee extensions, and others were performed while seated on a chair. Hip flexions, lateral leg raises, and repetitions of other exercises were performed standing upright behind the chair and holding the back of the chair for stability. To strengthen lower extremities, a fixed weight was placed on the ankle while participants performed strengthening exercises. Weights of 0.50, 0.75, 1.00, and 1.50 kg were used in accordance with each participant's strength level as the resistance progressively increased. The exercises performed using these ankle weights included seated knee flexion and extension and standing knee flexion and extensions. Exercises using a resistance band: Resistance bands were used to strengthen lower body. Lower body exercises included leg extension and hip flexion
  Arms: Group 2

SUMMARY:
Patients with liver cirrhosis have severe physical deconditioning. Aim: To compare between the effect of neuromuscular electric stimulation(NMES) and exercises (EX)on treatment of patients with liver cirrhosis.

DETAILED DESCRIPTION:
70 patients have been chosen from department of internal medicine, Cairo university hospitals, Egypt. 5 patients refused to participate .65 patients divided randomly into 2 groups. All the procedures were explained to patients.2 patients refused to sign informed consent and excluded from the study. 31 patients in group1 and 32 patients in group2. 1patients dropped in group1 and excluded from the study and two patients didn't continued the programmed treatment in group 2 and their data removed.

Thirty patients in each group signed an informed consent and complete the treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Positive for anti-HCV.
* Not under antiviral therapy at entry.
* Positive for chronic hepatitis or compensated cirrhosis.
* Negative for hepatitis B surface (HBs) antigen.
* Free of co-infection with HIV.
* Not pregnant.
* Systolic blood pressure of less than 180 mmHg or diastolic blood pressure of less than 110 mmHg.
* (viii)No ischemic heart disease or severe arrhythmia

Exclusion Criteria:

* Significant cardiac disease (ejection fraction <60% or history of coronary artery disease).
* Chronic renal failure on dialysis.
* Hemoglobin <11.0 g/L.
* Human immunodeficiency virus infection.
* Hepatocellular carcinoma.
* Active non-hepatocellular carcinoma related malignancy.
* Myopathy.
* Any physical impairment or orthopedic abnormality preventing EX, or post-liver transplantation

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Sitting standing test | 12 week
  number of cycle /30 seconds
Balance | 12 weeks
  Seconds
Time up and go test | 12 weeks
  number of cycle / minute
6 Minutes walk distance | 12 weeks
  distance walked in 6 minutes
2 Minutes steps test | 12 weeks
  number of steps in 2 minutes.
Chronic liver diseases questionnaire (CLDQ) | 12 week
  score
SF-36 | 12 week
  Score

CONTACTS AND LOCATIONS:
Overall Officials: Manal K Youssef, Principal Investigator — Cairo university, Egypt
Locations (1):
- Manal K. youssef, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data shared on reasonable request from corresponding author.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2 months
Access Criteria: reasonable request from corresponding author.